CLINICAL TRIAL: NCT01994304
Title: Assessment and Evaluation of the Safe Childbirth Checklist --Phase II Rajasthan, India
Brief Title: Assessment and Evaluation of the Safe Childbirth Checklist --Phase II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Foundation of India (Other)
Collaborators: UBS Optimus Foundation (Other); The Children's Investment Fund Foundation (Other)
Responsible Party: Principal Investigator, Dr. Beena Varghese, Sr. Health Economist and Additional Professor, Public Health Foundation of India
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SCC--P2
Record Dates: First submitted 2013-11-13; First posted 2013-11-25 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Intrapartum Mortality
Keywords: Safe Childbirth Checklist; Intrapartum mortality, Quality of Institutional delivery care; Maternal & newborn care practices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No safe childbirth checklist (No Intervention): The selected control districts include Bharatpur, Pali, Jhunjhunu, and Nagaur
- Safe Childbirth Checklist (Active Comparator): The selected districts for SCC intervention include Alwar, Jalore, Sirohi, Sikar, Dausa, and Churu
  Interventions: Behavioral: SCC

INTERVENTIONS:
Behavioral: SCC — The intervention involves introducing and orienting health providers on the SCC, facilitating availability of a specific set of commodities and regular targeted supervision. These are expected to improve adherence to life saving interventions immediately before, during and after birth, and reduce intrapartum mortality (still births and very early neonatal deaths).
  Arms: Safe Childbirth Checklist

SUMMARY:
PHFI independently evaluated the effectiveness of the Safe Childbirth Checklist program in preventing stillbirths and early neonatal deaths. Evaluation used a quasi-experimental design with data collection from 34 facilities across six intervention districts and four control districts. The study with a sample of 137,000 births has 88% power to detect 15% reduction in intrapartum mortality. Data on this was collected over a period of 17 months (November 2013 to April 2015).

DETAILED DESCRIPTION:
The Safe Childbirth Checklist (SCC), a tool that provides reminders and is a job aid to health care providers is a new maternal and newborn care intervention that is being implemented by the Government of Rajasthan with technical support from Jhpeigo. SCC is thus expected to improve the quality of delivery care practices and was implemented in Community Health Centres (CHCs) and District Hospitals (DHs) across seven districts in Rajasthan over a two-year time period (2013 to 2015). PHFI independently evaluated the effectiveness and cost-effectiveness of the SCC in preventing intrapartum (stillbirths and very early neonatal deaths within 3-days after births). Data on 137,000 births was collected over a period of 17 months (November 2013 to April 2015) from 34 facilities with sick newborn care centres (SNC).

Facility records were main source of outcome data. Labor room provided data on stillbirths whereas information on very early neonatal deaths came from SNCs. All Data collection and management was done through software specifically developed for this purpose.

For a better understanding on how maternal and neonatal complications are diagnosed and managed at the facility, in-depth interviews were conducted with the service providers (specialists, physicians, labor room staff nurses, and pharmacists) from the District hospitals and CHCs. In addition, interviews focused on understanding the use, acceptability and feasibility of the SCC among various types of providers.

Cost of this intervention was estimated from a program perspective, and cost effectiveness in terms of cost per perinatal death prevented was calculated.

Preliminary analysis has found that SCC is significantly associated with a 11% reduction in intrapartum deaths.

Permission for this study and data collection has been obtained from the Department of Health and Family Welfare, Government of Rajasthan.

ELIGIBILITY:
Inclusion Criteria:

* All women who deliver at the District Hospitals (DHs), Sub-District Hospitals (SDHs) and Community Health Centres (CHCs)

Exclusion Criteria:

-

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200000 (Actual)
Dates: Start 2012-06; Primary Completion 2015-09 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Perinatal mortality | 18 months (Nov-2013 to May-2015)
  This evaluation will independently estimate the effectiveness of the Safe Childbirth Checklist in reduce perinatal mortality by 15% in the intervention areas

SECONDARY OUTCOMES:
Morbidity rates for infants and mothers | 18 months (Nov-2013 to May-2015)
  We determine checklist-related morbidity rates for infants and mothers at the intervention facilities by observing the following:
  1. Level of Practices -use of partograph or recording of events; active management of third stage labor (AMTSL); early initiation of breast feeding; use of antihypertensives/magnesium sulphate for mothers and use of antibiotics for mother and neonate
  2. Levels of neonatal morbidity (low birth weight/prematurity, asphyxia, sepsis), maternal morbidity (Post partum haemorrhage, sepsis, eclampsia etc)

CONTACTS AND LOCATIONS:
Overall Officials: Beena Varghese, PhD, Principal Investigator — Public Health Foundation of India
Locations (1):
- Public Health Foundation of India, New Delhi, New Delhi, India

REFERENCES:
- [Derived] Varghese B, Copas A, Kumari S, Bandyopadhyay S, Sharma J, Saha S, Yadav V, Kumar S. Does the safe childbirth checklist (SCC) program save newborn lives? Evidence from a realistic quasi-experimental study, Rajasthan, India. Matern Health Neonatol Perinatol. 2019 Mar 1;5:3. doi: 10.1186/s40748-019-0098-4. eCollection 2019. PMID 30867935
- See also: Saving lives through checklist — http://ciff.org/impact/saving-babies-lives-rajasthan/